CLINICAL TRIAL: NCT04984304
Title: Individualized Diagnosis and Treatment of Extraesophageal Reflux in Patients With Chronic Cough
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNO-ENT-EER_Cough
Record Dates: First submitted 2021-06-01; First posted 2021-07-30 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Chronic Cough; Extraesophageal Reflux; Laryngopharyngeal Reflux; Allergy; Asthma
Keywords: chronic cough; extraesophageal reflux; laryngopharyngeal reflux; allergy; asthma
MeSH Terms: conditions — Chronic Cough; Laryngopharyngeal Reflux; Hypersensitivity; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mild cough (Experimental): Mild cough only slightly worsening the quality of life (VAS 1-3)
  Interventions: Behavioral: Lifestyle modifications and Antireflux diet
- Moderate and severe cough (Experimental): Moderate and severe cough that significantly worsen the quality of life (VAS 4-10)
  Interventions: Diagnostic Test: Extraesophageal reflux diagnostic

INTERVENTIONS:
Behavioral: Lifestyle modifications and Antireflux diet — Patients in Arm 1 - mild cough only slightly worsening the quality of life (VAS 1-3) will undergo treatment using lifestyle modifications and an Antireflux diet for 3 months.
  Arms: Mild cough
Diagnostic Test: Extraesophageal reflux diagnostic — Patients in Arm 2 - moderate and severe cough that significantly worsen the quality of life (VAS 4-10) will undergo extraesophageal reflux diagnostics consisting of esophageal 24-hour pH/Impedance Reflux Monitoring and peptest study on fasting
  Arms: Moderate and severe cough

SUMMARY:
Chronic cough is a very unpleasant symptom, significantly reduces the patient's quality of life, and bothers the neighborhood. A very common cause or co-factor of chronic cough is extraesophageal reflux (EER).

The aim of the project is the precise diagnosis of EER in patients with chronic cough (in patients with a simultaneously diagnosed allergic cause and without it).

DETAILED DESCRIPTION:
Chronic cough is a very unpleasant symptom, significantly reduces the patient's quality of life, and bothers the neighborhood. A very common cause or co-factor of chronic cough is extraesophageal reflux (EER). Liquid reflux, or even just aerosol reflux, causes mucosal inflammation and sensitizes the mucous membrane of the airways, which is then sensitive to even slight noxa. The cough then further damages the mucosa, creating a vicious circle. EER can be the main cause of chronic cough, but also a worsening cofactor of cough in patients with other causes (allergic and non-allergic bronchial asthma, chronic rhinosinusitis, and others).

The aim of the project is the precise diagnosis of EER in patients with chronic cough (in patients with a simultaneously diagnosed allergic cause and without it). Accurate diagnosis and assessment of severity allow patients to be divided into 2 groups. The group with mild symptoms and the findings will be treated in the first phase with diet and lifestyle modifications. With a positive response to this "conservative" type of treatment, patients would not have to undergo a series of tests. Patients with severe problems and confirmed EER will be treated individually according to recommended measures.

Study protocol

* signing of Informed Consent
* anamnestic questionnaire (age, sex, weight, height, smoking, alcohol, reflux disease, treatment of allergic disease, pyrosis, treatment of reflux disease)

Allergology examination

* Cough Visual Analogue Scale (VAS)
* Hull Airway Reflux Questionnaire
* Asthma Control Test
* Spirometry
* Prick Tests
* Fractional Exhaled nitric oxide (FeNO) test
* Laboratory tests (IgE, specific IgE, ECP)

Otorhinolaryngologic examination

* Cough Visual Analogue Scale (VAS)
* RSS -12 (Reflux Symptom Score - 12)
* RSA - Short version (Reflux Sign Assessment - Short version)
* The Perceived Stress Scale
* Evaluation of Compliance with Antireflux Precaution Visual Analogue Scale (VAS)
* dividing patients into 2 arms

Arm 1 - mild cough only slightly worsening the quality of life (VAS 1-3) - treatment using lifestyle modifications and Antireflux diet for 3 months. In case of persistent severity of cough or worsening - continue to Arm 2 Arm 2 - moderate and severe cough that significantly worsen the quality of life (VAS 4-10)

Extraesophageal reflux diagnostic

* Esophageal 24-hour pH/Impedance Reflux Monitoring
* Peptest study on fasting

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years
* patients with chronic cough (cough that lasts 3 months or longer)
* consent with participation in the study

Exclusion Criteria:

* patients using ACE inhibitors or Angiotensin II receptor blockers
* patients with head and neck cancer
* patients after radiotherapy in the head and neck area
* patients with airway or lung cancer
* patients with chronic lung disease except for bronchial asthma (COPD, interstitial lung disease, bronchiectasis, respiratory bronchiolitis)
* patients with chronic rhinosinusitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
EER severity and type and allergy | 6 months
  Comparison of extraesophageal reflux severity and type in patients with chronic cough with or without concomitant allergic cause of cough. The number of EER events on impedance and improvement of RSA - Short version scale (Reflux Sign Assessment - Short version) will be observed and compared with improvement of objective measurements and clinical findings.

SECONDARY OUTCOMES:
Diet and life-style modifications and asthma | 6 months
  Evaluation of the importance of diet and life-style modifications in patients with mild symptoms findings of extraesophageal reflux in patients with concomitant bronchial asthma and without concomitant bronchial asthma. The percentage of recommended diet compliance will be compared with the scores of improvement of RSA - Short version scale (Reflux Sign Assessment - Short version) and clinical findings.
Allergic diseases and chronic cough with concomitant extraesophageal reflux | 6 months
  Comparison of the frequency of individual allergic diseases in patients with chronic cough and concomitant extraesophageal reflux.
Individual phenotypes of bronchial asthma in patients with EER | 6 months
  Comparison of the frequency of individual phenotypes of bronchial asthma in patients with proven extraesophageal reflux.
Asthma severity and control | 6 months
  Evaluation of the evolution of asthma severity and the level of asthma control in patients with bronchial asthma and extraesophageal reflux while following a diet and life-style modifications. The percentage of recommended diet compliance will be correlated with the possibility to discontinue administration of selected drugs (e.g. corticosteroids and biological treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Viktória Hránková, MD,PhD,FESO, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kahrilas PJ, Altman KW, Chang AB, Field SK, Harding SM, Lane AP, Lim K, McGarvey L, Smith J, Irwin RS; CHEST Expert Cough Panel. Chronic Cough Due to Gastroesophageal Reflux in Adults: CHEST Guideline and Expert Panel Report. Chest. 2016 Dec;150(6):1341-1360. doi: 10.1016/j.chest.2016.08.1458. Epub 2016 Sep 7. PMID 27614002
- [Background] Kanemitsu Y, Kurokawa R, Takeda N, Takemura M, Fukumitsu K, Asano T, Yap J, Suzuki M, Fukuda S, Ohkubo H, Maeno K, Ito Y, Oguri T, Niimi A. Clinical impact of gastroesophageal reflux disease in patients with subacute/chronic cough. Allergol Int. 2019 Oct;68(4):478-485. doi: 10.1016/j.alit.2019.04.011. Epub 2019 Jun 7. PMID 31182314
- [Background] Shirai T, Mikamo M, Tsuchiya T, Shishido Y, Akita T, Morita S, Asada K, Fujii M, Suda T. Real-world effect of gastroesophageal reflux disease on cough-related quality of life and disease status in asthma and COPD. Allergol Int. 2015 Jan;64(1):79-83. doi: 10.1016/j.alit.2014.08.001. Epub 2014 Oct 22. PMID 25605530
- [Background] Herregods TVK, Pauwels A, Jafari J, Sifrim D, Bredenoord AJ, Tack J, Smout AJPM. Determinants of reflux-induced chronic cough. Gut. 2017 Dec;66(12):2057-2062. doi: 10.1136/gutjnl-2017-313721. Epub 2017 Mar 15. PMID 28298354